CLINICAL TRIAL: NCT00494832
Title: Influence of Dexmedetomidine on the Evoked Potentials During Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31416-A; 064705 A01 (Other: University of Washington)
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Spine Surgery
Keywords: Dexmedetomidine; Evoked potentials; Spine surgery
MeSH Terms: interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine infusion
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Normal Saline infusion
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — 10 minutes loading dose of 0.9 mcg/kg
  Maintenance dose of 0.6 mcg/kg/hour
  Other Names: Dexmedetomidine hydrochloride
  Arms: Dexmedetomidine
Drug: Normal Saline — 10 minutes loading dose of 0.9 mcg/kg
  Maintenance dose of 0.6 mcg/kg/hour
  Other Names: 0.9% Sodium Chloride
  Arms: Placebo

SUMMARY:
The purposes of this study are:

1. To evaluate the safety and efficacy of Dexmedetomidine as an adjunct for anesthesia during spine surgery and
2. To investigate the influence of Dexmedetomidine on the evoked potentials.

DETAILED DESCRIPTION:
Use of evoked potentials can significantly improve neurologic outcome after major spine surgery. Modalities of evoked potentials commonly used are Somato-Sensory Evoked Potentials (SSEP's), Motor Evoked Potentials (MEP's), and Visual Evoked Potentials (VEP's).

Dexmedetomidine (DEX) is an alpha-2 agonist and has been FDA approved as an adjunct sedative agent to general anesthesia. It has been purported to reduce the amount of anesthetic required and potentiate the analgesic effect of opiates. In addition, DEX was shown to have minimal effect on SSEP's and VEP's in both rats and humans. Any decrease in the dose of general anesthesia that improves the monitoring of evoked potentials, supports DEX as an adjunct.

It is known that all anesthetic agents can interfere with the recording of evoked potentials. The choice of anesthetic however, depends on the modality of neurophysiologic monitoring planned for the patient. Total intravenous anesthesia (TIVA) and Sevoflurane, a low dose inhalational anesthetic are the usual agents for spine surgery. Both have a dose-related depressant effect on the quality of evoked potentials. As a result, it is common practice for the anesthesiologist to adjust the depth of anesthesia to improve signaling. The use of either anesthetic must accompany continuous infusion of Propofol and an opioid, Remifentanil or Fentanyl. The anesthesiologist then decides whether DEX should be as an adjunct. In our experience, DEX did not impair evoked potentials. In fact, it improved the quality of signals in a few patients. Yet, there are no published data of such effects in medical literature.

We hypothesize that Dexmedetomidine will not influence evoked potentials when used as an adjunct to general anesthesia. Our study is prospective, randomized, double-blinded and will be carried out on a set of anesthetics. We will first evaluate DEX as an adjunct in TIVA, then as an adjunct to Sevoflurane. The probable benefit of DEX may avoid the use of potent inhaled anesthetics which would improve VEP's monitoring. Quality recording of evoked potentials can enhance our ability to detect iatrogenic injury to the spinal cord and vision.

ELIGIBILITY:
Inclusion Criteria:

* Adult spine surgery patients requiring evoked potentials monitoring.

Exclusion Criteria:

* Age younger than 18 and older than 80 years
* Patients with moderate neurological deficit
* ASA grade above 3
* Any chronic psychiatric disorder
* Body mass index (BMI) above 35
* Patients with cortical blindness, cataracts, retinal or optic neuropathy, glaucoma, untreated diabetes, active hepatitis, active coronary artery disease, untreated arrhythmias and patients with renal or hepatic insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in evoked potentials | Duration of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Irene Rozet, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Rozet I, Metzner J, Brown M, Treggiari MM, Slimp JC, Kinney G, Sharma D, Lee LA, Vavilala MS. Dexmedetomidine Does Not Affect Evoked Potentials During Spine Surgery. Anesth Analg. 2015 Aug;121(2):492-501. doi: 10.1213/ANE.0000000000000840. PMID 26097987